CLINICAL TRIAL: NCT00481676
Title: A Randomized, 24 Weeks, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Assess the Efficacy and Safety of Omalizumab in Adult Patients With Chronic Urticaria Who Exhibit IgE Against Thyroperoxidase
Brief Title: Efficacy and Safety of Omalizumab in Adults (18-70 Years) With Moderate to Severe Chronic Urticaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIGE025ADE05
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Results first posted 2011-10-21 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2011-09

CONDITIONS: Chronic Urticaria
Keywords: Chronic urticaria, omalizumab, thyroperoxidase, IgE
MeSH Terms: conditions — Chronic Urticaria; Epilepsy, Idiopathic Generalized | interventions — Omalizumab; Loratadine; Clemastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omalizumab 75-375 mg (Experimental): Omalizumab was dosed at 75 to 375 mg according to baseline IgE and body weight as described in dosing tables in the study protocol. Dosing occurred subcutaneously every 2 or 4 weeks depending on dose.
  Interventions: Drug: Omalizumab 75-375 mg; Drug: Loratadine
- Placebo to omalizumab (Placebo Comparator): Placebo to omalizumab was dosed at 75 to 375 mg according to baseline IgE and body weight as described in dosing tables in the study protocol. Dosing occurred subcutaneously every 2 or 4 weeks depending on dose.
  Interventions: Drug: Placebo to omalizumab; Drug: Loratadine; Drug: Clemastine

INTERVENTIONS:
Drug: Omalizumab 75-375 mg — Omalizumab was supplied as lyophilized, sterile powder in a single-use, 5 ml vial designed to deliver 150 mg of omalizumab upon reconstitution with 1.4 ml sterile water for injection.
  Other Names: Xolair
  Arms: Omalizumab 75-375 mg
Drug: Placebo to omalizumab — Placebo to omalizumab was supplied as lyophilized, sterile powder in a single-use, 5 ml vial designed to deliver 150 mg placebo to omalizumab upon reconstitution with 1.4 ml sterile water for injection.
  Arms: Placebo to omalizumab
Drug: Loratadine — All participants received antihistamines on demand (loratadine and clemastine), as the trial was designed to investigate the effect of omalizumab as an add-on to antihistamines in people with chronic urticaria (CU). Administration of antihistamines is the current gold standard treatment of CU. A significant proportion of people with CU is not well controlled by this standard or by using high doses of antihistamines.
  Other Names: Lorano®
Drug: Clemastine — All participants received antihistamines on demand (loratadine and clemastine), as the trial was designed to investigate the effect of omalizumab as an add-on to antihistamines in people with chronic urticaria (CU). Administration of antihistamines is the current gold standard treatment of CU. A significant proportion of people with CU is not well controlled by this standard or by using high doses of antihistamines.
  Other Names: Tavegil®
  Arms: Placebo to omalizumab

SUMMARY:
This study evaluated the safety and efficacy of omalizumab in adult patients with moderate to severe chronic urticaria who exhibit IgE against thyroperoxidase.

ELIGIBILITY:
Inclusion criteria:

* Males or females from 18-70 years of age
* Body weight ≥ 20 kg and ≤ 150 kg and with a total serum IgE level ≥ 30 IU/mL and ≤ 700 IU/mL
* Specific serum IgE anti-TPO level ≥ 8.0 IU/mL, documented within 3 months prior to randomization or time of pre-screening
* Diagnosis of moderate to severe chronic urticaria
* Subject's current episode of chronic urticaria according to the European Academy of Allergology and Clinical Immunology/Global Allergy and Asthma European Network/European Dermatology Forum (EAACI/GA2LEN/EDF) guideline at the time of screening
* Current episode of chronic urticaria has not responded to the approved marketed dose of antihistamine for 2 weeks or longer
* Urticaria activity score (UAS) ≥ 0 at any of the 7 days of the first section of the screening period
* UAS7 ≥ 10 at the time of randomization

Exclusion criteria:

* Females of child-bearing potential or breast feeding
* Present or past medical conditions that could have interfered with the study results
* Randomized into any other omalizumab study or who had received omalizumab
* Received investigational drugs within 30 days of enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- Germany (11):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Giessen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Munich

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omalizumab 75-375 mg | Placebo to Omalizumab
Started | 27 | 22
Completed | 25 | 17
Not Completed | 2 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Unsatisfactory therapeutic effect | 1 | 4
Not completed — Administrative problem | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab 75-375 mg | Placebo to Omalizumab | Total
Number analyzed (Participants) | 27 | 22 | 49
Age Continuous [Mean (Standard Deviation); unit: years] | 39.1 (9.0) | 42.3 (15.0) | 40.5 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 8 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in the Weekly Urticaria Activity Score (UAS7) From Baseline to the End of the Study (Week 24)
Description: The UAS is a composite diary-recorded score with numeric severity ratings (0=none to 3=intense) for the number of wheals per 24 hours and the intensity of the pruritus. The total daily score (sum of the wheal and pruritus scores) ranges from 0 to 6. Because of variations in chronic urticaria disease intensity, assessment of disease activity was based on a weekly (7 days) UAS score called UAS7, that is, the sum of the daily UASs, ranging from 0 to 42 per week. A higher score indicates worse disease. A negative change score (Week 24 score minus Baseline score) indicates improvement.
Time Frame: Baseline to end of the study (Week 24)
Population: Intent-to-treat (ITT) population: All randomized patients who received at least 1 dose of study drug and had at least 1 post-baseline assessment of the primary efficacy variable.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Omalizumab 75-375 mg | Placebo to Omalizumab
Number analyzed (Participants) | 27 | 22
Units on a scale | -17.8 (10.52) | -5.8 (11.52)

2. Secondary Outcome: Number of Patients With Wheals, Erythemas, Pruritus, and Angioedemas at the End of the Study
Description: Patients kept a daily diary of the number of wheals and erythema and the severity of pruritus and angioedemas during the study.
Time Frame: At the end of the study (Week 24)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Omalizumab 75-375 mg | Placebo to Omalizumab
Number analyzed (Participants) | 27 | 22
Participants
  Wheals - None | 19 | 1
  Wheals - < 10 | 3 | 11
  Wheals - 10-50 | 1 | 3
  Wheals - > 50 | 1 | 1
  Erythemas - None | 18 | 4
  Erythemas - < 10 | 4 | 7
  Erythemas - 10-50 | 1 | 4
  Erythemas - > 50 | 1 | 1
  Pruritus - None | 16 | 2
  Pruritus - Mild | 4 | 8
  Pruritus - Moderate | 3 | 3
  Pruritus - Severe | 1 | 3
  Angioedema - None | 21 | 8
  Angioedema - Mild | 1 | 6
  Angioedema - Moderate | 0 | 1
  Angioedema - Severe | 2 | 1

3. Secondary Outcome: Standardized (With Respect to Length of Time) Area Under the Curve (AUC) for the Urticaria Activity Score (UAS) From Baseline to the End of the Study (Week 24)
Description: The UAS is a composite diary-recorded score with numeric severity ratings (0=none to 3=intense) for the number of wheals per 24 hours and the intensity of the pruritus. The total daily score (sum of the wheal and pruritus scores) ranges from 0 to 6. A higher score indicates worse disease. AUC was calculated from daily UASs where no urticaria medication was taken using the trapezoidal rule. The standardized AUC UAS was calculated as the sum of trapezoids divided by the length of time.
Time Frame: Baseline to the end of the study (Week 24)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Omalizumab 75-375 mg | Placebo to Omalizumab
Number analyzed (Participants) | 27 | 21
Units on a scale | 1.0 (1.28) | 2.5 (1.23)

4. Secondary Outcome: Use of Concomitant and Rescue Medications
Description: Data was collected from the patients' diaries about the number of clemastine and loratadine pills taken during the last 7 days of each month of the study.
Time Frame: At Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Pills
Arm/Group | Omalizumab 75-375 mg | Placebo to Omalizumab
Number analyzed (Participants) | 27 | 22
Pills
  Week 4 - clemastine (N=27,21) | 0.7 (3.10) | 3.7 (5.30)
  Week 4 - loratadine (N=27,22) | 1.3 (2.51) | 4.2 (2.61)
  Week 8 - clemastine (N=26,20) | 1.3 (4.05) | 2.4 (3.69)
  Week 8 - loratadine (N=26,21) | 1.2 (2.45) | 4.2 (2.62)
  Week 12 - clemastine (N=25,17) | 1.1 (3.81) | 1.8 (3.80)
  Week 12 - loratadine (N=25,19) | 1.2 (2.33) | 3.3 (2.64)
  Week 16 - clemastine (N=24,16) | 0.2 (0.72) | 1.4 (2.13)
  Week 16 - loratadine (N=24,17) | 0.6 (1.56) | 3.6 (3.00)
  Week 20 - clemastine (N=24,16) | 0.9 (3.88) | 2.2 (2.88)
  Week 20 - loratadine (N=24,17) | 0.5 (1.47) | 4.6 (3.48)
  Week 24 - clemastine (N=23,14) | 0.7 (2.72) | 1.4 (2.13)
  Week 24 - clemastine (N=23,16) | 0.3 (1.11) | 3.3 (2.50)

5. Secondary Outcome: Change in the Dermatology Life Quality Index (DLQI) Score From Baseline to the End of the Study (Week 24)
Description: The DLQI is a dermatology-specific quality of life (QoL) questionnaire designed for use in patients over 16 years of age. Patients are asked to respond to each of 10 questions on a 4-point Likert scale in regard to how much their skin problem has affected their life over the last week (0=not at all, 1=a little, 2=a lot, 3=very much). The overall (total) DLQI score (range=0 to 30) is calculated by summing the scores of all 10 questions. The higher the score, the more QoL is impaired. A negative change score (Week 24 score minus Baseline score) indicates improvement.
Time Frame: Baseline to the end of the study (Week 24)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Omalizumab 75-375 mg | Placebo to Omalizumab
Number analyzed (Participants) | 27 | 22
Units on a scale
  Baseline (N=27, 22) | 10.1 (6.04) | 9.8 (5.29)
  Week 24 (N=27,21) | 3.7 (7.12) | 8.1 (6.11)
  Week 24 minus Baseline (N=27,21) | -6.3 (8.36) | -1.5 (5.83)

6. Secondary Outcome: Change in the Skindex Score From Baseline to the End of the Study (Week 24)
Description: Skindex is a 30-item questionnaire with 3 scores (functioning, emotions,symptoms) and a composite score (average scale score) that assesses the effects of skin disease on patients' quality of life (QoL). Item responses are standardized on a scale from 0 to 100. The mean of all 61 items was calculated. A higher score indicates a lower QoL. A negative change score (Week 24 score minus Baseline score) indicates improvement.
Time Frame: Baseline to the end of the study (Week 24)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Omalizumab 75-375 mg | Placebo to Omalizumab
Number analyzed (Participants) | 27 | 22
Units on a scale
  Baseline (N=27,22) | 1.8 (0.69) | 1.6 (0.53)
  Week 24 (N=27,21) | 0.9 (1.00) | 1.5 (0.79)
  Week 24 minus Baseline (N=27,21) | -0.9 (0.89) | -0.1 (0.61)

7. Secondary Outcome: Change in Chronic Urticaria Quality of Life (CU-Q2oL) Scores From Baseline to the End of the Study (Week 24)
Description: The CU-Q2oL (German version) is a questionnaire that measures the relative burden of chronic urticaria on subjective well-being. It has 23 questions in 3 domains (symptoms, general impairment, difficulties and problems due to urticaria). Patients are asked to respond how much they are troubled by each problem on a 5-point Likert scale (1=not at all to 5=very much). Each domain and the overall (total) scores are normalized to a scale of 1 to 100. A higher score indicates lower QoL. A negative change score (Week 24 score minus Baseline score) indicates improvement.
Time Frame: Baseline to the end of the study (Week 24)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Omalizumab 75-375 mg | Placebo to Omalizumab
Number analyzed (Participants) | 27 | 22
Units on a scale
  Baseline : Limits Looks (N=27,21) | 31.5 (23.86) | 34.5 (24.97)
  Baseline : Swelling/eating (N=27,22) | 21.8 (20.17) | 26.7 (19.97)
  Baseline : Sleep (N=27,22) | 45.8 (24.02) | 46.6 (23.91)
  Baseline : Mental status (N=27,22) | 42.6 (21.72) | 42.4 (18.71)
  Baseline : Functioning (N=27,22) | 36.0 (22.47) | 30.7 (15.88)
  Baseline : Itching/embarrassment (N=27,22) | 58.1 (18.97) | 56.8 (14.80)
  Baseline : Total score (N=27,22) | 39.5 (16.34) | 38.9 (8.87)
  Week 24 : Limits looks (N=27,21) | 17.1 (20.26) | 23.2 (20.27)
  Week 24 : Swelling/eating (N=27,21) | 10.4 (23.58) | 27.4 (23.92)
  Week 24 : Sleep (N=27,21) | 27.3 (29.73) | 47.3 (27.36)
  Week 24 : Mental status (N=27,21) | 25.9 (27.77) | 40.1 (25.22)
  Week 24 : Functioning (N=27,21) | 11.9 (22.43) | 27.0 (20.73)
  Week 24 : Itching/embarrassment (N=27,21) | 22.9 (29.42) | 57.4 (22.41)
  Week 24 : Total score (N=27,21) | 18.5 (22.66) | 37.3 (16.22)
  Week 24 - Baseline: Limits looks (N=27,20) | -14.4 (24.69) | -9.4 (18.08)
  Week 24 - Baseline: Swelling/eating (N=27,21) | -11.3 (22.40) | -0.6 (18.74)
  Week 24 - Baseline: Sleep (N=27,21) | -18.5 (27.05) | -0.6 (23.13)
  Week 24 - Baseline: Mental status (N=27,21) | -16.7 (27.35) | -2.4 (19.57)
  Week 24 - Baseline: Functioning (N=27,21) | -24.1 (23.94) | -3.8 (21.08)
  Week 24 - Baseline: itching/embarrassmen (N=27,21) | -35.2 (32.71) | -0.9 (20.76)
  Week 24 - Baseline: Total score (N=27,21) | -21.0 (21.97) | -2.3 (14.14)

8. Secondary Outcome: Patient's Global Assessment of Their Chronic Urticaria Symptoms
Description: Patients made a global assessment of their chronic urticaria symptoms on a 4-point Likert scale (none, mild moderate, severe) at Baseline and again at the end of the study. The number of patients in each category is reported.
Time Frame: At Baseline and at the end of the study (Week 24)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Omalizumab 75-375 mg | Placebo to Omalizumab
Number analyzed (Participants) | 27 | 22
Participants
  Baseline: Missing | 0 | 0
  Baseline: No complaints | 3 | 0
  Baseline: Moderate complaints | 13 | 13
  Baseline: Severe complaints | 11 | 8
  Baseline: Maximum complaints | 0 | 1
  Week 24: Missing | 1 | 1
  Week 24: No complaints | 16 | 3
  Week 24: Moderate complaints | 6 | 7
  Week 24: Severe complaints | 3 | 9
  Week 24: Maximum complaints | 1 | 2

9. Secondary Outcome: Investigator's Global Assessment of the Patient's Chronic Urticaria Symptoms
Description: The investigator made a global assessment of the patient's chronic urticaria symptoms on a 4-point Likert scale (none, mild, moderate, severe) at Baseline and again at the end of the study. The number of patients in each category is reported.
Time Frame: At Baseline and at the end of the study (Week 24)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Omalizumab 75-375 mg | Placebo to Omalizumab
Number analyzed (Participants) | 27 | 22
Participants
  Baseline: Missing | 1 | 0
  Baseline: None | 1 | 0
  Baseline: Mild | 7 | 9
  Baseline: Moderate | 13 | 6
  Baseline: Severe | 5 | 7
  Week 24: Missing | 0 | 1
  Week 24: None | 18 | 1
  Week 24: Mild | 6 | 9
  Week 24: Moderate | 1 | 4
  Week 24: Severe | 2 | 7

ADVERSE EVENTS:
Arm/Group | Omalizumab 75-375 mg | Placebo to Omalizumab
Serious Adverse Events (participants affected / at risk) | 0/27 | 2/22
Other Adverse Events (participants affected / at risk) | 19/27 | 12/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab 75-375 mg (N=27) | Placebo to Omalizumab (N=22)
Eye Infection (Infections and infestations) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab 75-375 mg (N=27) | Placebo to Omalizumab (N=22)
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Injection Site Pain (General disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Gastrointestinal Infection (Infections and infestations) | 3 | 2
Nasopharyngitis (Infections and infestations) | 9 | 11
Sinusitis (Infections and infestations) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Headache (Nervous system disorders) | 10 | 6
Insomnia (Psychiatric disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 3
Eczema (Skin and subcutaneous tissue disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. any publications from a single-site are postponed until the publication of the pooled date (ie, data from all sites) in the clinical trial.